CLINICAL TRIAL: NCT00874822
Title: Prevalence of Sleep Apnea in Patients Presenting for Hip or Knee Replacement Surgery
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0212-09-EP
Record Dates: First submitted 2009-03-26; First posted 2009-04-03 (Estimated); Results first posted 2012-01-20 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Berlin: Patients diagnosed with obstructive sleep apnea by polysomnography after being screened with the Berlin questionnaire.

SUMMARY:
The study hypothesis is that the prevalence of obstructive sleep apnea in patients presenting for total knee or total hip arthroplasty is higher than generally suspected. The study will include just one arm and results will be compared to a literature control group. Participants referred for preoperative evaluation will be screened using a standard questionnaire. Those at high risk of obstructive sleep apnea will then undergo a formal overnight sleep study (polysomnography).

DETAILED DESCRIPTION:
The study hypothesis is that the prevalence of obstructive sleep apnea in patients presenting for total knee or total hip arthroplasty is higher than generally suspected. The study will include just one arm and results will be compared to a literature control group, a study performed by Harrison et al. and published in the December 2003 issue of The Journal of Arthroplasty. Participants referred for preoperative evaluation will be screened using a standard questionnaire. Those at high risk of obstructive sleep apnea will then undergo a formal overnight sleep study (polysomnography). The Berlin questionnaire is being used for screening.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Planned total hip or total knee arthroplasty
* Referral to the internal medicine preoperative evaluation clinic

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are all patients referred to an academic internal medicicine preoperative evaluation clinic prior to hip or knee arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2009-05-26 (Actual); Primary Completion 2012-04-11 (Actual); Study Completion 2012-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason F Shiffermiller, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Kaw R, Michota F, Jaffer A, Ghamande S, Auckley D, Golish J. Unrecognized sleep apnea in the surgical patient: implications for the perioperative setting. Chest. 2006 Jan;129(1):198-205. doi: 10.1378/chest.129.1.198. PMID 16424433
- [Background] Ancoli-Israel S, Kripke DF, Klauber MR, Mason WJ, Fell R, Kaplan O. Sleep-disordered breathing in community-dwelling elderly. Sleep. 1991 Dec;14(6):486-95. doi: 10.1093/sleep/14.6.486. PMID 1798880
- [Background] Young T, Evans L, Finn L, Palta M. Estimation of the clinically diagnosed proportion of sleep apnea syndrome in middle-aged men and women. Sleep. 1997 Sep;20(9):705-6. doi: 10.1093/sleep/20.9.705. PMID 9406321
- [Background] Gupta RM, Parvizi J, Hanssen AD, Gay PC. Postoperative complications in patients with obstructive sleep apnea syndrome undergoing hip or knee replacement: a case-control study. Mayo Clin Proc. 2001 Sep;76(9):897-905. doi: 10.4065/76.9.897. PMID 11560300
- [Background] Harrison MM, Childs A, Carson PE. Incidence of undiagnosed sleep apnea in patients scheduled for elective total joint arthroplasty. J Arthroplasty. 2003 Dec;18(8):1044-7. doi: 10.1016/s0883-5403(03)00459-5. PMID 14658110

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Berlin
Started | 216
Completed | 208
Not Completed | 8
Not completed — excluded by criteria | 8

BASELINE CHARACTERISTICS:
Arm/Group | Berlin
Number analyzed (Participants) | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 99
  >=65 years | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.88 (0.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 98
Region of Enrollment [Number; unit: participants]
  United States | 216

OUTCOME MEASURES:

1. Primary Outcome: Obstructive Sleep Apnea
Description: The number patients with obstructive sleep apnea whether newly diagnosed or known at study entry.
Time Frame: 9 Months
Measure: Number; unit: participants
Arm/Group | Berlin
Number analyzed (Participants) | 216
participants | 41
Statistical Analysis 1: Comparison: Berlin; Ho: The Prevalence of obstructive sleep apnea in patients planning hip or knee arthroplasty will be no different using current screening techniques than it was in a historical control group. The prevalence of OSA in the study population is hypothesized to be at least 10% higher than the best previous estimate of 6.7%. Employing a two-sided hypothesis test with α of 0.05 and power of 0.85 yields a sample size of 163; Test type: Superiority or Other; p < 0.0001, Chi-squared, Corrected; Percentage of Participants = 19, 95% CI 2-sided [13.6 to 24.4], Standard Error of Mean 2.7

ADVERSE EVENTS:
Time Frame: 9 months
Description: Serious and other (nonserious) adverse events were not collected.
Arm/Group | Berlin
All-Cause Mortality (participants affected / at risk) | 0/216
Serious Adverse Events (participants affected / at risk) | 0/216
Other Adverse Events (participants affected / at risk) | 0/216

LIMITATIONS AND CAVEATS:
Obstructive sleep apnea was diagnosed in only four patients due to a high rate of failure to undergo PSG by patients for whom it was indicated. A second major weakness is the use of a literature control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes